CLINICAL TRIAL: NCT06255067
Title: "Efficacy of Noisome as A Carrier of Locally Delivered Minocycline Hydrochloride Gel in Stage II or Stage III Periodontitis: A Randomized Controlled Clinical Trial With Biochemical Analysis"
Brief Title: Efficacy of Noisome as A Carrier of Locally Delivered Minocycline Hydrochloride Gel
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, israa saiid, MSc student, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FDASU-RecIM022002
Record Dates: First submitted 2023-12-26; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Periodontitis
Keywords: Minocycline hydrochloride
MeSH Terms: conditions — Periodontitis; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Minocycline hydrochloride with noisome as carrier (Experimental): Group I ( Minocycline hydrochloride with noisome carrier)
  15 patients will receive the drug ( Minocycline hydrochloride with noisome carrier gel) at intervals 1,3,7&14 days
  Interventions: Drug: Minocycline hydrochloride with noisome carrier
- Minocycline hydrochoride only (Active Comparator): Group II (Minocycline hydrochloride only)
  15 patients will receive the drug (Minocycline hydrochloride only gel) at intervals 1,3,7&14 days
  Interventions: Drug: Minocycline Hydrochloride only

INTERVENTIONS:
Drug: Minocycline hydrochloride with noisome carrier — patient will receive Non-surgical debridement followed by injection of local delivery drug in the deepest pocket site, This will be done one day, three days, seven days and fourteen days
  Arms: Minocycline hydrochloride with noisome as carrier
Drug: Minocycline Hydrochloride only — patient will receive Non-surgical debridement followed by injection of local delivery drug in the deepest pocket site, This will be done one day, three days, seven days and fourteen days
  Arms: Minocycline hydrochoride only

SUMMARY:
The goal of this clinical trial is to compare the efficacy of Noisome as carrier of minocycline hydrochloride gel to minocycline hydrochloride in Stage II or Stage III Periodontitis . The main questions it aims to answer are:

* Is the Noisome carrier of minocycline hydrochloride has an effect in comparing to minocycline hydrochloride in Stage II or Stage III Periodontitis?
* what is the release profile of of minocycline hydrochloride noisome gel and minocycline hydrochloride gel? Participants will be asked to maintain oral hygiene after application of treatment Researchers will compare the effect of noisome as a carrier of locally delivered minocycline hydrochloride gel to minocycline hydrochloride gel in stage II or stage III periodontitis patients as an adjunct to non-surgical periodontal treatment] to see if Plaque Index (PI) , Gingival index,Clinical attachment level (CAL) &Periodontal Pocket Depth decreased or not.

DETAILED DESCRIPTION:
This study is designed to be a Randomized, Controlled, blinded, clinical trial; the eligible participants will be randomly allocated for one of the two comparative parallel-Groups; test and control group . The interventions will be prepared by the pharmacist and coded and the whole-time frame for the study will be 18 weeks.

The intervention to all participants will be Non-surgical debridement the the test group will receive the Noisome minocycline hydrochloride & control group will receive minocycline hydrochloride.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing to commit for the entire period of the trial and agreed to sign the written consent after full explanation of the study.
* Generalized Periodontitis (Stage II or stage III ) Patients; ( ≥ 3 mm CAL, PD 5-7 mm ) , premolar-molar area (test site) .
* Having more than 16 tooth excluding wisdom and test teeth that still had both mesial and distal neighboring teeth.
* Systemically free according to the modified Burkitt's health history questionnaire

Exclusion Criteria:

* Non-surgical periodontal therapy within the previous 12 months, systemic or local use of antibiotics with the previous 3 months, medication with possible influence on the periodontium.
* Pregnancy or contraceptives usage.
* Breastfeeding.
* Known allergy to the ingredients of the treatment.
* Smokers.
* vulnerable group; prisoners & orphans .

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-25 (Estimated); Primary Completion 2024-05-25 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
To measure clinical assessment Plaque Index (PI) in both groups (mincycline hydrochloride with noisome as carrier & minocycline hydrochloride only) | measured at the baseline, before the application of drug& after 18 weeks
  To measure the clinical parameter Plaque Index (PI) on score from zero to three
  0 = No plaque in gingival area.
  1. = A film of plaque adhering to the free gingival margin and adjacent area of tooth. The plaque may be recognized only by running a probe across the tooth surface.
  2. = Moderate accumulation of soft deposit within the gingival pocket and on the gingival pocket and on the gingival margin and/or adjacent tooth surface that can be seen by naked eye.
  3. = Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface.
To measure clinical assessment Gingival Index (GI) in both groups (mincycline hydrochloride with noisome as carrier & minocycline hydrochloride only) | measured at the baseline, before the application of drug& after 18 weeks
  To measure the clinical parameter gingival Index(GI) on score from zero to three
  Gingival index (GI) 0 = Normal gingiva.
  1. = Mild inflammation, slight change in color, slight edema; no bleeding on probing.
  2. = Moderate inflammation, redness, edema, and glazing; bleeding on probing.
  3. = Sever inflammation, marked redness and edema, ulceration; tendency to spontaneous bleeding.
To measure Clinical attachment level (CAL) in both groups (mincycline hydrochloride with noisome as carrier & minocycline hydrochloride only) | measured at the baseline, before the application of drug& after 18 weeks
  To measure Clinical attachment level (CAL) in millimeter (mm).
To measure Periodontal Pocket Depth (PPD) in both groups (mincycline hydrochloride with noisome as carrier & minocycline hydrochloride only) | measured at the baseline, before the application of drug& after 18 weeks
  To measure Periodontal Pocket Depth (PPD) in millimeter (mm).

SECONDARY OUTCOMES:
- Evaluate the releasing profile of minocycline hydrochloride noisome gel and minocycline hydrochloride gel | first day then third day then seventh day lastly after fourteen days
  change in number of releasing profile of each drug

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Fouad, PHD, Study Director — AinShams University
Locations (1):
- AinShams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
sharing the inclusion& exclusion criteria , study design, intervention ,statistical data &references.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Jain R, Mohamed F, Hemalatha M. Minocycline containing local drug delivery system in the management of chronic periodontitis: A randomized controlled trial. J Indian Soc Periodontol. 2012 Apr;16(2):179-83. doi: 10.4103/0972-124X.99259. PMID 23055582
- [Background] Apatzidou DA, Kinane DF. Nonsurgical mechanical treatment strategies for periodontal disease. Dent Clin North Am. 2010 Jan;54(1):1-12. doi: 10.1016/j.cden.2009.08.006. PMID 20103469
- [Background] Cortelli JR, Querido SM, Aquino DR, Ricardo LH, Pallos D. Longitudinal clinical evaluation of adjunct minocycline in the treatment of chronic periodontitis. J Periodontol. 2006 Feb;77(2):161-6. doi: 10.1902/jop.2006.040409. PMID 16460239
- [Background] Nakao R, Takigawa S, Sugano N, Koshi R, Ito K, Watanabe H, Senpuku H. Impact of minocycline ointment for periodontal treatment of oral bacteria. Jpn J Infect Dis. 2011;64(2):156-60. PMID 21519133
- [Background] Uchegbu IF, Vyas SP (2015). Non-Ionic surfactant based vesicles (noisome) in drug delivery. Int J Pharm. ;172:33-70.
- [Background] Williams RC, Paquette DW, Offenbacher S, Adams DF, Armitage GC, Bray K, Caton J, Cochran DL, Drisko CH, Fiorellini JP, Giannobile WV, Grossi S, Guerrero DM, Johnson GK, Lamster IB, Magnusson I, Oringer RJ, Persson GR, Van Dyke TE, Wolff LF, Santucci EA, Rodda BE, Lessem J. Treatment of periodontitis by local administration of minocycline microspheres: a controlled trial. J Periodontol. 2001 Nov;72(11):1535-44. doi: 10.1902/jop.2001.72.11.1535. PMID 11759865